CLINICAL TRIAL: NCT03776227
Title: A Bioequivalence Study Testing Two Formulations of Sotagliflozin in Healthy Male and Female Subjects Under Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BEQ14993; U1111-1205-3319 (Other: UTN)
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus; Healthy Subjects
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sotagliflozin Test (Experimental): One tablet of sotagliflozin administered orally under fasting conditions
  Interventions: Drug: sotagliflozin (SAR439954)
- Sotagliflozin Reference (Active Comparator): Two tablets of sotagliflozin administered orally under fasting conditions
  Interventions: Drug: sotagliflozin (SAR439954)

INTERVENTIONS:
Drug: sotagliflozin (SAR439954) — Pharmaceutical form: tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

To determine the bioequivalence of a single dose of one tablet of sotagliflozin (test) compared to two tablets of sotagliflozin (reference) under fasting conditions in healthy male and female subjects

Secondary Objectives:

* To evaluate the single-dose pharmacokinetics of sotagliflozin following administration of one tablet sotagliflozin (test) compared to two tablets of sotagliflozin (reference) in healthy male and female subjects under fasting conditions
* To evaluate safety and tolerability of one tablet sotagliflozin (test) compared to two tablets of sotagliflozin (reference) administered under fasted conditions in healthy male and female subjects

DETAILED DESCRIPTION:
Study duration per participant is approximately 103 days including a screening period up to 21 days before first dose, 4 periods of dosing and pharmacokinetic (PK) sampling each lasting 7 days, a washout period of 8-21 days between dosing, and an end of study visit 10-15 days after the last dose.

ELIGIBILITY:
Inclusion criteria :

* Healthy male or female subjects, between 18 and 55 years of age, inclusive.
* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female.
* Body mass index between 18.0 and 30.0 kg/m2, inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs after 10 minutes resting in supine position and after 3 minutes in standing position:

  * 95 mmHg < systolic blood pressure (SBP) <140 mmHg
  * 45 mmHg < diastolic blood pressure (DBP) <90 mmHg
  * 40 bpm < heart rate (HR) <100 bpm
* Standard 12-lead electrocardiogram (ECG) parameters after 10 minutes resting in supine position in the following ranges; 120 ms<PR<220 ms, QRS<120 ms, QTc≤430 ms if male, ≤450 ms if female and normal ECG tracing unless the Investigator considers an ECG tracing abnormality to be not clinically relevant.
* Laboratory parameters within the normal range, unless the Investigator considers an abnormality to be clinically irrelevant for healthy subjects; however serum creatinine, alkaline phosphatase, hepatic enzymes (aspartate aminotransferase, alanine aminotransferase), and total bilirubin (unless the subject has documented Gilbert syndrome) should not exceed the upper laboratory norm.
* Female subject must use a double contraception method including a highly effective method of birth control, except if she has undergone sterilization at least 3 months earlier or is postmenopausal. The accepted double contraception methods include the use of 2 of the following 3 contraceptive options: (1) intrauterine device; (2) hormonal contraception; (3) condom or diaphragm or cervical/vault cap, in addition to spermicide. Menopause is defined as being amenorrheic for at least 2 years with plasma follicule-stimulating hormone (FSH) level >30 UI/L. Hormonal contraception is acceptable in this study (contraceptive guidance will be described in the study protocol).
* Having given written informed consent prior to undertaking any study-related procedure.
* Not under any administrative or legal supervision.
* Male subject, whose partners are of childbearing potential (including lactating women), must accept to use, during sexual intercourse, a double contraception method according to the following algorithm: (condom) plus (intra-uterine device or hormonal contraceptive) from the inclusion up to 3 months after the last dosing. Male subject, whose partners are pregnant, must use, during sexual intercourse, a condom from the inclusion up to 3 months after the last dosing.
* Male subject has agreed not to donate sperm from the inclusion up to 3 months after the last dosing.

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal (especially pancreatitis), hepatic (especially biliary disease, including cholecystectomy), renal, metabolic, hematological, neurological, musculoskeletal, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* History of renal disease, or significantly abnormal kidney function test (glomerular filtration rate (GFR) <90 mL/min as calculated using the Cockcroft-Gault equation (7) at screening.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Blood donation of a pint or more within 2 months before inclusion.
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 3 minutes when changing from supine to standing position.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day on a regular basis).
* Smoking more than 5 cigarettes or equivalent per day and/or unable to stop smoking during the study.
* Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day).
* If female, pregnancy (defined as positive human chorionic gonadotropin (β-HCG blood test), breast-feeding.
* Any medication (over-the counter or prescription medications, including St John's Wort), or any herbal supplements or supra-therapeutic vitamins within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the substance; any vaccination within the last 28 days, and any biologics (antibody or its derivatives) given within 4 months before inclusion.
* Any subject who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Any subject in the exclusion period of a previous study according to applicable regulations.
* Any subject who cannot be contacted in case of emergency.
* Any subject who is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti hepatitis C virus antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti HIV1 and anti HIV2 Ab).
* Positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
* Positive alcohol test.
* Any consumption of citrus (grapefruit, orange, etc) or their juices within 5 days before inclusion.
* Any history or presence of deep leg vein thrombosis or pulmonary embolism or a recurrent or frequent history of deep vein thrombosis in first degree relatives (parents, siblings or children).
* Any presence or history of urinary tract infection or genital mycotic infection in the last 4 weeks before screening.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1 of each period
  Maximum plasma concentration observed
AUC 0-72h (area under the curve) | Day 1 to Day 3 of each period
  Truncated AUC 0-72h

SECONDARY OUTCOMES:
Time to reach Cmax (tmax) | Day 1 of each period
  Time to reach Cmax
Terminal half-life (t1/2z) | Day 1 to Day 7 of each period
  Terminal half-life associated with the terminal slope (λz)
Area under the plasma concentration versus time curve (AUClast) | Day 1 to Day 7 of each period
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time tlast
Adverse events | Day 1 to Day 7 of each period
  Number of participants with adverse events
Electrocardiograms (ECGs) | Day 1 to Day 7 of each period
  Number of patients with clinically significant changes in electrocardiograms (ECGs)
Vital signs | Day 1 to Day 7 of each period
  Number of patients with clinically significant changes in vital signs
Clinical laboratory tests | Day 1 to Day 7 of each period
  Number of patients with clinically significant changes in clinical laboratory tests
Area under the curve (AUC) | Day 1 to Day 7 of each period
  Area under the plasma concentration versus time curve extrapolated to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 8400001, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org